CLINICAL TRIAL: NCT05409209
Title: Carotid Plaque Length to Predict Cardiovascular Events
Status: Active, not recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Putuo Hospital, Shanghai University of Traditional Chinese Medicine (Unknown); 904th Hospital of the Joint Logistics Support Force of the PLA (Other); Gongli Hospital (Unknown); Yueyang Hospital, Shanghai University of Traditional Chinese medicine (Unknown)
Responsible Party: Principal Investigator, Pan Li, Clinical Professor, Changhai Hospital
Other Study IDs: CPLi-2017
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease
Keywords: Carotid Artery Ultrasound; Carotid Plaque; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Carotid plaque length: Patients underwent carotid ultrasonography and first coronary angiography simultaneously

SUMMARY:
This multicenter study involved 5 hospitals (Changhai Hospital; Yueyang Hospital of Shanghai University of Traditional Chinese Medicine; Gongli Hospital; Putuo Hospital of Shanghai University of Traditional Chinese Medicine; No. 904 Hospital of the PLA Joint Logistics Support Force Wuxi). The study enrolled 3000 patients for suspected CAD who referred to coronary angiography from January 2017 through December 2018.

DETAILED DESCRIPTION:
Patients with coronary artery disease who were confirmed by coronary angiography were eligible for the study. Carotid ultrasonography was performed before coronary angiography, and carotid intima-media thickness (IMT), maximum thickness and length of all plaques were measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients≥18 years old, those who underwent carotid ultrasonography and first coronary angiography simultaneously.

Exclusion Criteria:

* Patients with known coronary artery disease, previous coronary or carotid revascularization, missing carotid ultrasound or coronary angiography results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for first coronary angiography and underwent carotid ultrasonography simultaneously
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
major cardiovascular event | 3 years
  A composite of cardiovascular death, myocardial infarction, and ischemic stroke

SECONDARY OUTCOMES:
major vascular event | 3 years
  A composite of cardiovascular death, myocardial infarction, ischemic stroke, and coronary artery revascularization
all-cause death | 3 years
cardiovascular death | 3 years
myocardial infarction | 3 years
ischemic stroke | 3 years
coronary artery revascularization | 3 years
  coronary artery bypass grafting or percutaneous coronary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pan Li, PhD, Principal Investigator — Changhai Hospital; Jian Na, MD, Study Director — Putuo Hospital; Liang Chen, MD, Study Director — 904th Hospital of the Joint Logistics Support Force of the PLA; Wei Zhang, MD, Study Director — Gongli Hospital; Yawei Yang, MD, Study Director — Yueyang Hospital
Locations (5):
- China (5):
  - No. 904 Hospital of the PLA Joint Logistics Support Force, Wuxi, Jiangsu
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Gongli Hospital, Shanghai, Shanghai Municipality
  - Putuo Hospital, Shanghai, Shanghai Municipality
  - Yueyang Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided